CLINICAL TRIAL: NCT05564936
Title: The ME&MG Digital Solution for Autonomous Assessment of Myasthenia Gravis: a Validation Study
Brief Title: The ME&MG Digital Solution for Autonomous Assessment of Myasthenia Gravis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ad scientiam (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DOMYA
Record Dates: First submitted 2022-09-27; First posted 2022-10-04 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- MG patients (Experimental): MG patients will perform 3 in-clinic visits and use the ME&MG app at-home during 12 months
  Interventions: Device: ME&MG mobile application
- Healthy volunteers (Other): Healthy volunteers will perform one in-clinic visit and will use the app at-home once
  Interventions: Device: ME&MG mobile application

INTERVENTIONS:
Device: ME&MG mobile application — ME&MG is a standalone software (digital solution) running on patients smartphones, connected to a web portal for physicians. It is intended to be used as an unsupervised digital self-assessment tool for the monitoring of disabilities in patients living with MG.

SUMMARY:
ME&MG is a standalone software (digital solution) running on patients smartphones, connected to a web portal for physicians. It is intended to be used as an unsupervised digital self-assessment tool for the monitoring of disabilities in patients living with MG.

ME&MG contains digital active tests for the assessment of ptosis, breathing, dysarthria, upper- and lower-limb (arms and legs) weakness, treatment follow-up, and validated e-questionnaires related to daily activities, pain, fatigue, sleep, and depression disorders.

The objectives of this study are to validate the accuracy, reliability and reproducibility of the unsupervised at-home self-assessment of symptoms on the patient's smartphone with ME&MG versus the standard in-clinic testing, as well as to evaluate the safety of the solution, its usability and satisfaction.

DETAILED DESCRIPTION:
Myasthenia gravis (MG) is an autoimmune neuromuscular disease characterised by fatigable muscle weakness due to autoantibodies targeting components of the neuromuscular junction.

Deficits are measured using validated clinical scales such as the Quantitative Myasthenia Gravis score (QMG) QMG, Myasthenia Gravis Composite Score (MCS), Myasthenia Gravis Activities of Daily Living score (MG-ADL), etc., Unfortunately, this type of assessment might require expensive material, time, and personnel training, which make MG assessment difficult for clinicians in routine care.

Research on the matter has highlighted the importance of Patient-Reported Outcomes (PROs), composite measures of disease severity and quality-of-life measurements. This has led to the development of a number of tools for the self-assessment of PROs with validated questionnaires. However, there is no tool that overcomes the constraints of standard tests such as the QMG while allowing for the collection of objective data and PROs between visits.

ME&MG is a standalone software (digital solution) running on patients smartphones, connected to a web portal for physicians. It is intended to be used as an unsupervised digital self-assessment tool for the monitoring of disabilities in patients living with MG.

ME&MG contains digital active tests for the assessment of ptosis, breathing, dysarthria, upper- and lower-limb (arms and legs) weakness, treatment follow-up, and validated e-questionnaires related to daily activities, pain, fatigue, sleep, and depression disorders.

The objectives of this study are to validate the accuracy, reliability and reproducibility of the unsupervised at-home self-assessment of symptoms on the patient's smartphone with ME&MG versus the standard in-clinic testing, as well as to evaluate the safety of the solution, its usability and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 Years
* Diagnosed with gMG at screening with generalized muscle weakness meeting the clinical criteria for diagnosis of MG, as defined by the MGFA Clinical Classification Class II, III, or IV, and likely not in need of a respirator for the duration of the study, as judged by the investigator
* With positive serologic testing for anti-AChR autoantibody at screening
* Have read the information sheet and signed the informed consent form
* Own a personal smartphone which software version is above 13 for IOS and 8 for Android included
* Able to use a smartphone
* Able to read language in which the mobile application is available (French, English, Spanish) and able to understand pictograms

Exclusion Criteria:

* Subjects having undergone thymectomy Plasma Exchange Therapy or Intravenous Immunoglobulin Therapy within four weeks of screening
* Subjects having initiated FcRn inhibitor therapy within the four weeks preceding screening
* Known medical or psychological condition(s) or risk factor(s) that, as judged by the investigator, might interfere with the subject's full participation in the study, pose any additional risk for the subject, or confound the assessment of the subject or outcome of the study.
* Pregnant and nursing women
* Person under guardianship or curatorship
* Current drugs or/and alcohol abuse that could influence performance on the tests, as judged by the investigator
* Participant included in another ME&MG clinical study
* Participant has participated in another clinical study within the previous 30 days of screening or is currently participating in another study that, in the opinion of the Investigator, might interfere with the subject's full participation in the study or confound the assessment of the subject or outcome of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2025-09-24 (Estimated); Study Completion 2026-09-24 (Estimated)

PRIMARY OUTCOMES:
To demonstrate that ME&MG tests results performed at-home, under unsupervised condition, are correlated to standard tests results performed in-clinic, under supervised conditions | baseline
  Pearson correlation coefficient will be used to assess the relationship between digital tests versus standard tests

SECONDARY OUTCOMES:
To compare results between in-clinic digital tests and in-clinic standard tests, test to test | baseline
  pearson correlation coefficient between digital tests and standard tests
To assess reproducibility between in-clinic digital tests and at-home digital tests | baseline, day 1, day 89, day 90
  intraclass correlation coefficient
To assess test-retest reliability of at-home digital tests | Day1, Day 2, Day 3, Day 87, Day 88, Day 89
  intraclass correlation coefficient mean k raters (ICCk; k=day)
To compare results obtained with the at-home ME&MG composite score and the in-clinic standard QMG composite score | baseline, day 1
  Pearson correlation coefficient between digital composite score and QMG score
To assess adverse events related to the use of the mobile application | through study completion, an average of 1 year
  Descriptive analysis of adverse events (AEs) related to the use of the application
To assess satisfaction and user experience with the smartphone application | through study completion, an average of 1 year
  descriptive analysis of questionnaires resulsts
To assess correlation of the at-home ME&MG composite score with the Myasthenia Gravis Activities of Daily Living (MG-ADL) score | baseline, day 90, day 365
  Pearson's correlation coefficient between ME&MG composite score and MG-ADL scores
to assess daily activites | 12 months
  Myasthenia Gravis Activities of Daily Living (MG-ADL)
to assess depression | 12 months
  Patient Health Questionnaire-8 (PHQ8)
to assess pain | 12 months
  pain likert scale
to assess insomnia | 12 months
  Insomnia Severity Index
To assess at-home compliance to the ME&MG smartphone application | through study completion, an average of 1 year
  descriptive analysis of adherence data
To assess quality of life | Baseline, day 90, Day 365
  36-Item Short Form Survey (SF-36)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (11):
  - University of Colorado Denver, Aurora, Colorado
  - University of Florida Health, Jacksonville, Florida
  - HealthParterns Institute, Bloomington, Indiana
  - Indiana University Health, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Neurological Associates of Long Island, P.C., Lake Success, New York
  - Duke University, Durham, North Carolina
  - OHSU, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - The University of Tennessee Medical Center, Knoxville, Tennessee
  - Vanderbilt Health, Nashville, Tennessee
- France (8):
  - Hôpital Raymond Poincaré, Garches
  - CHU Grenoble, Grenoble
  - Hôpital Salengro, Lille
  - CHRU Nancy, Nancy
  - CHU Nantes, Nantes
  - Pitié-Salpêtrière, Paris
  - CHU de Strasbourg - Hôpital de Hautepierre, Strasbourg
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No